CLINICAL TRIAL: NCT04872816
Title: Study of the Effect of Obstructive Sleep Apnea on Telomere Length and Its Associated Mechanisms
Brief Title: Obstructive Sleep Apnea and Telomere Length
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Prof. Dr. Lia Azeredo-Bittencourt, Clinical Professor, Associação Fundo de Incentivo à Pesquisa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0232/2018
Record Dates: First submitted 2021-04-26; First posted 2021-05-05 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep; Telomere; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous airway positive pressure (Experimental): All participants in continuous airway positive pressure arm will use CPAP (model S10-Resmed®) with expiratory relief and nasal mask.
  Interventions: Device: Continuous airway positive pressure
- SHAM continuous airway positive pressure (Sham Comparator): Individuals in SHAM continuous airway positive pressure arm will use CPAP (model S7-Resmed®) with expiratory relief and nasal mask. The Sham-CPAP consists of a modified CPAP so that the pressure in the mask was less than 1 cm H2O. In this study, the Sham-CPAP equipment includes an increase in the expiratory orifice of the CPAP mask to eliminate airflow resistance, and a resistor with a small orifice was placed between the CPAP and the circuit. The noise produced by the ventilator and the airflow through the mask will be very similar to that of the effective CPAP. The diameter of the expiratory orifice was 10 cm H2O, and a 4 mm diameter resistor was placed between the trachea and the CPAP flow generator.
  Interventions: Device: Continuous airway positive pressure

INTERVENTIONS:
Device: Continuous airway positive pressure — The continuous airway positive pressure will be used as the gold-standard treatment for obstructive sleep apnea for 6 months

SUMMARY:
Obstructive sleep apnea (OSA) is a highly prevalent and morbid sleep disorder. Among the factors associated with its pathophysiology, the role of intermittent hypoxia stands out, contributing to the development of oxidative stress and inflammation. It is known that cumulative levels of these factors negatively influence the final portion of the DNA, known as telomere. In this sense, the investigators hypothesize that OSA is capable of accelerating aging process through telomere shortening mediated by inflammatory and oxidative markers. Thus, the aim of this study is to investigate the effect of OSA and its treatment with CPAP on the variation of telomere length and their associated mechanisms. For this, a randomized, double-blind, sham-controlled clinical study with 6 months duration will be conducted. We will recruit male participants with OSA diagnosis (apnea-hypopnea indexe15/hour), aged between 35-65 years and body mass index<35 kg/m2, which will be randomized to use CPAP or sham-CPAP for 6 months. Participants will visit the laboratory 7 times (baseline and after 1, 2, 3, 4, 5 and 6 months) and will be submitted to clinical and otorhinolaryngological evaluation, sleep questionnaires, polysomnography and blood collection for DNA and extraction and measurement of telomere length, as well as the expression of telomerase and oxidative and inflammatory markers (ADMA, homocysteine, cysteine, TBARS, 8-oxodG, TNF-a, IL-6 and IL-10). This project aims to contribute to the elucidation of the effect of OSA on telomere length maintenance, as well as the adjacent mechanisms to this relationship.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) of less than 35kg/m2
* age between 35 and 65 years
* diagnosed by laboratory polysomnography with moderate to severe OSA (apnea-hypopnea index, AHI≥20 events/hour of sleep)

Exclusion Criteria:

* illiteracy
* participants with more than 50% of the respiratory events obtained in the polysomnography exam being central apneas
* participants with central AHI>5 events/hour of sleep
* participants with sleepiness, measured by the Epworth sleepiness scale≥14
* participants with severe otorhinolaryngological diseases that preclude the use of CPAP (severe nasal septum deviation, severe nasal turbinate hypertrophy, marked palatine and/or adenoid hypertrophy)
* abuse of alcohol or chronic use of psychoactive drugs
* participants with decompensated clinical, neurological or psychiatric illness
* participants with other sleep disorders; participants who had already undergone previous OSA treatments

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change of Leukocyte telomere length from baseline to 6 months | 6 months
  It will be evaluated the change between leukocyte telomere length before and after the intervention

SECONDARY OUTCOMES:
Change of sleep quality assessed by Pittsburgh Sleep Quality index from baseline to 6 months | 6 months
  It will be evaluated the change between sleep quality before and after the intervention

OTHER OUTCOMES:
Change of depressive symptoms assessed by Beck depression inventory from baseline to 6 months | 6 months
  It will be evaluated the change between depressive symptoms before and after the intervention
Change of body mass index from baseline to 6 months | 6 months
  It will be evaluated the change between body mass index before and after the intervention
Change of anxiety symptoms assessed by Anxiety status scale from baseline to 6 months | 6 months
  It will be evaluated the change between anxiety symptoms before and after the intervention
Change of cervical circumference from baseline to 6 months | 6 months
  It will be evaluated the change between cervical circumference before and after the intervention
Change of abdominal circumference from baseline to 6 months | 6 months
  It will be evaluated the change between abdominal circumference before and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No